CLINICAL TRIAL: NCT06378554
Title: Cereset Research for Performance Improvement in a Hospital Nursing Unit
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: The Susanne Marcus Collins Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00111227
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Health Personnel; Stress; Anxiety; Insomnia; Depression
Keywords: Anxiety; Stress; Insomnia; Cereset Research; Brain electrical activity; Neurotechnology; HIRREM; Neuromodulation; Acoustic stimulation; Healthcare Worker
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Cereset Intervention Group (Active Comparator): This system uses the same core technology and algorithms to echo brainwaves in real-time using audible tones, as with High-resolution, relational, resonance-based, electroencephalic mirroring (HIRREM).
  Interventions: Device: Cereset Research
- No Intervention (No Intervention): No Intervention

INTERVENTIONS:
Device: Cereset Research — The upgraded platform for medical research using the HIRREM technology has been rebranded as Cereset Research® (CR). This system uses the same core technology and algorithms to echo brainwaves in real-time using audible tones, as with High-resolution, relational, resonance-based, electroencephalic mirroring (HIRREM). The CR system also includes 64-bit processing architecture for faster feedback, the use of 4 sensors, and the use of standard protocols (with flexibility regarding the length and sequencing of the standard protocols), all done with eyes closed. Four sensors are applied to the scalp at a time. However, only two sensors are actively echoing feedback. The software automatically switches from one sensor pair to the other when needed. This reduces the number of sensor placement changes needed, resulting in shorter session time and fewer interruptions.
  Arms: Cereset Intervention Group

SUMMARY:
The purpose of this study is to explore whether an implementation process composed of offering CR to staff in a single hospital nursing unit has any potential impact on unit-level quality measures post-implementation.

DETAILED DESCRIPTION:
This is a pre-post design quality improvement project and implementation study, evaluating implementation measures, group level quality measures using QI methodology, and individual-level behavioral and performance measures before and after implementation of the Cereset Research (CR) evidence-based intervention among nursing unit staff. Individual-level behavioral symptoms and a nursing performance metric will be evaluated among healthcare workers in the nursing unit in the pre- and post-implementation timeframes among individuals who consent to participate in these evaluation activities. Up to 40 members of the unit will have the opportunity to enroll in the acoustic echoing neurostimulation intervention during the implementation timeframe. The neurostimulation intervention consists of 4 Cereset Research sessions of audible tones echoing current brainwave activity, and individual level behavioral symptoms will be collected following the last intervention session.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comply with basic instructions and be able to sit still, comfortably during sessions.
* Healthcare worker in the Orthopedic Trauma Unit at Atrium Health Wake Forest Baptist, aged 18 years and older.

Exclusion Criteria:

* Unable, unwilling, or incompetent to provide informed consent.
* Physically unable to come to the study visits.
* Severe hearing impairment (because CR involves acoustic stimulation that participants would need to be able to hear).
* Weight is over the chair limit (400 pounds).
* Currently enrolled in another Cereset Research study.
* Use of the following modalities within one month before enrollment: electroconvulsive therapy (ECT), prior use of transcranial magnetic stimulation (TMS), transcranial direct current stimulation (TDCS), alpha stimulation, eye movement desensitization and reprocessing (EMDR), brain spotting, neurofeedback, biofeedback, or deep brain stimulation (DBS). Individuals will be given the opportunity to discontinue these techniques for one month and then enroll.
* Known seizure disorder.
* Thoughts of active suicide within the last 3 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percent of ortho trauma unit staff who complete Cereset intervention | up to 2 years
  Percent of ortho trauma unit staff who complete CR Intervention

CONTACTS AND LOCATIONS:
Overall Officials: Charles H Tegeler, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No